CLINICAL TRIAL: NCT03305393
Title: Implementation of a Protocol Utilizing Adaptive CRT in a Normal AV Conduction, CRT Non-Response Population at Generator Replacement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Only one subject was enrolled and that subject was Lost to Follow Up. Decision was made to terminate the study.
Sponsor: Stern Cardiovascular Foundation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMPROVE RESPONSE
Record Dates: First submitted 2017-08-15; First posted 2017-10-10 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Heart Failure
Keywords: Heart Failure; CRT; Cardiac Recynchronization Therapy; left bundle branch block; atrio-ventricular conduction
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Adaptiv CRT (Other): Adaptiv CRT algorithm in Medtronic FDA approved CRT devices to be programmed as ON at 6 month follow-up visit
  Interventions: Device: Adaptiv CRT

INTERVENTIONS:
Device: Adaptiv CRT — Adaptiv CRT algorithm to be programmed to ON in CRT devices of study patients at 6 month follow-up visit

SUMMARY:
IMPROVE RESPONSE is a physician initiated research study. It is a prospective, non-randomized, multi-center, post-market, U.S. Cardiac Resynchronization Therapy (CRT) in heart failure (HF) observational study. The purpose of this clinical study is to test the hypothesis that market-released CRT devices, which contain the AdaptivCRT (aCRT) algorithm have an incremental benefit in improving CRT response in a chronic CRT non responder population with left bundle branch block (LBBB) and normal atrio-ventricular (AV) condition compared to CRT devices with traditional biventricular pacing delivery methods at generator replacement.

ELIGIBILITY:
Inclusion Criteria:

* Normal AV conduction (SAV<220 ms or PAV<270 MS)
* Left Bundle Branch Block (defined as > or = to 140 ms (male) or > or = 130 (female), QR or rS in leads V1 and V2, and Mid QRS notching or slurring in v 2 of leads V1, V2, V5, V6 and I and aVL.)
* Patient and/or physician assessment or unchanged or worsened heart failure status at the time of recommended replacement time (RRT) for previous CRT device.
* Sinus Rhythm at the time of enrollment

Exclusion Criteria:

* Moderate to severe Aortic Stenosis
* Moderate to severe Mitral Regurgitation
* Patient age <18 years old
* AF burden >15%
* Severe pulmonary disease requiring supplemental oxygen use
* ESRD
* System Modification at RRT Generator Changeout
* AdaptivCRT prior to enrollment
* Expected patient longevity < 1 year
* Persistant or chronic atrial fibriliation
* Women who are pregnant or who plan to become pregnant during the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-06-11 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
Ejection fraction | 12 Months
  Change in ejection fraction as determined by echocardiography 6 months following the addition of adaptive CRT as compared to the same end points following patient management optimization
NYHA functional class | 12 months
  Change in NYHA functional class 6 months following the addition of adaptive CRT as compared to the same end points following patient management optimization

SECONDARY OUTCOMES:
Atrial fibrillation burden | 12 Months
  Atrial fibrillation burden and/or progression to permanent atrial fibrillation as determined by device interrogation and review
Heart failure hospitalizations | 12 months
  Amount and severity of heart failure hospitalizations and health care utilization as reported by subjects
Left ventricular end systolic volume | 12 months
  As determined by echocardiographic evidence
Time to first appropriate therapy for VT and/or VF | 12 months
  Time determined by device interrogation from sensing to response
Percentage of RV synchronized LV pacing | 12 months
  Percentage determined by device interrogation and compared to clinical outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Stern Cardiovascular Foundation, Germantown, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No